CLINICAL TRIAL: NCT03528018
Title: Efficacy of a Combined Transcranial Direct Current Stimulation and Virtual Reality-based Paradigm for Upper Limb Rehabilitation in Individuals With Severe Hemiparesia. A Randomized Control Trial Survivor With Severe Hemiparesis
Brief Title: Efficacy of a Combined Transcranial Direct Current Stimulation and Virtual Reality Intervention
Acronym: REACT01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospitales Nisa (Other)
Collaborators: Universitat Politècnica de València (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NISA-PHYS-2016/1; TIN2014-61975-EXP (Other Grant/Funding Number: Ministerio de Economía y Competitividad of Spain); BES-2014-068218 (Other Grant/Funding Number: Ministerio de Economía y Competitividad of Spain)
Record Dates: First submitted 2018-04-24; First posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Stroke; Hemiparesis; Chronic Stroke; Upper Limb Injury
Keywords: Virtual Reality; Rehabilitation; Physical therapy
MeSH Terms: conditions — Stroke; Paresis; Arm Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Conventional physical therapy
  Interventions: Other: Physical therapy
- Experimental (Experimental): Combined tDCS and VR-based intervention
  Interventions: Device: REACt system; Other: Physical therapy

INTERVENTIONS:
Device: REACt system — The REACt system is a virtual reality-based paradigm for upper limb rehabilitation that allows for interaction of individuals with restricted movements from active responses triggered when they attempt to perform a movement. The experimental system also provides multisensory stimulation in the visual, auditory, and tactile channels, and transcranial direct current stimulation coherent to the observed movements
  Arms: Experimental
Other: Physical therapy — Physical therapy included passive and active mobilization of the paretic upper limb. Passive range of motion exercises were provided in those segments where no active movement was detected to meticulously reproduce a range of articular movements and muscle and soft tissue elongation. In case of residual active movement capability, participants were encouraged to perform the movements with the assistance of the therapists

SUMMARY:
Rehabilitation options for stroke survivors who present severe hemiparesis in chronic stages are limited and may end in compensation techniques that involve the use of the less affected arm to achieve some degree of functional independence. Transcranial direct current stimulation (tDCS) is a non-invasive technique that has been used after stroke to promote excitability of the surviving neural architecture in order to support functional recovery. Interestingly, cortical excitability has been reported to increase when tDCS is combined with virtual reality. This synergetic effect could explain the promising results achieved by preliminary experimental interventions that combined both approaches on upper limb rehabilitation after stroke. The objective of this study is to explore the use of these interventions in subjects with severe hemiparesis and to determine its efficacy in comparison to conventional physical therapy

ELIGIBILITY:
Inclusion Criteria:

* chronicity > six months
* severe paresis of the upper limb defined by the Brunnstrom Approach as stages I or II and by the Upper Extremity subscale of the Fugl-Meyer Assessment as scores below 19
* ability to maintain a sitting position for at least 60 minutes
* fairly good cognitive condition defined by scores in the Mini-Mental State Examination above 23.

Exclusion Criteria:

* pacemakers
* brain implants or other metallic objects (valves, coils, etc.)
* impaired comprehension that hinder sufficient understanding of the instructions defined by Mississippi Aphasia Screening Test scores below 45
* severe visual impairments
* emotional or behavioral circumstances that impede adequate collaboration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2016-09-17 (Actual)

PRIMARY OUTCOMES:
Change in the Upper Extremity subscale of the Fugl-Meyer Assessment Scale from baseline to the end of the intervention and from the end of the intervention to one-month after the intervention | Pre-intervention (within 5 days prior intervention), post-intervention (within 5 days after intervention), one-month follow-up (within 30 to 35 days after the intervention)
  The Fugl-Meyer Assessment of Motor Recovery after Stroke evaluates and measures recovery in post-stroke hemiplegic patients in both clinical and research settings. Score range: 0-66

SECONDARY OUTCOMES:
Change in the Time subscale of the Wolf Motor Function Test from baseline to the end of the intervention and from the end to one-month after the intervention | Pre-intervention (within 5 days prior intervention), post-intervention (within 5 days after intervention), one-month follow-up (within 30 to 35 days after the intervention)
  The Wolf Motor Function Test is a quantitative measure of upper extremity motor ability through timed and functional tasks. Score range: 0-1200
Change in the Functional ability subscale of the Wolf Motor Function Test from baseline to the end of the intervention and from the end to one-month after the intervention. | Pre-intervention (within 5 days prior intervention), post-intervention (within 5 days after intervention), one-month follow-up (within 30 to 35 days after the intervention)
  The Wolf Motor Function Test is a quantitative measure of upper extremity motor ability through timed and functional tasks. Score range: 0-75
Change in the Nottingham Sensory Assessment from baseline to the end of the intervention and from the end to one-month after the intervention. | Pre-intervention (within 5 days prior intervention), post-intervention (within 5 days after intervention), one-month follow-up (within 30 to 35 days after the intervention)
  The Nottingham Sensory Assessment is a multi-modal sensory examination that includes tests of tactile sensation (Score range: 0-2) (light, touch, touch localization, temperature discrimination, pinprick sensation, bilateral simultaneous stimulation), kinesthesia (Score range:0-3), and stereognosis (Score range: 0-2)
Intrinsic Motivation Inventory | Post-intervention (within 5 days after intervention)
  The Intrinsic Motivation Inventory is a multidimensional questionnaire structured into various subscales. In this study, this questionnaire was used to assess participant interest/enjoyment, perceived competence, pressure/tension, and value/usefulness measures. Score range for each subscale: 1-7
System Usability Scale | Post-intervention (within 5 days after intervention)
  The System Usability Scale is a simple ten-item scale that serves as a global assessment of subjective usability. Score range: 0-100

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Llorens, PhD, Principal Investigator — Universitat Politècnica de València
Locations (1):
- Servicio de Neurorrehabilitación y Daño Cerebral de los Hospitales NISA, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No